CLINICAL TRIAL: NCT05983393
Title: Effect of Ultrasound-guided Bilateral Erector Spina Plan Block for Postoperative Analgesia in Patients Undergoing Multilevel Posterior Spinal Instrumentation.
Brief Title: Erector Spina Plane Block for Multilevel Major Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Gökçe Gişi, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/12-04
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Pain; Post Operative Pain
Keywords: Pain; postoperative analgesia; Erector spinae plane block; posterior spinal instrumentation
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): No block was performed
  Interventions: Procedure: Control
- Erector spinae plane block (Active Comparator): Erector spinae plane block was performed, morphine was administered with patient-controlled analgesia (PCA) and all patients were followed in the ward.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — Erector spinae plane block was performed
  Arms: Erector spinae plane block
Procedure: Control — Erector spinae plane block was not applied.
  Arms: Control group

SUMMARY:
Erector spinae plane (ESP) block is an interfacial plane block with visceral and somatic analgesic activity at paraspinal muscles. This study aims to examine the postoperative analgesic efficacy of ESP block in patients undergoing posterior spinal instrumentation

DETAILED DESCRIPTION:
Postoperative patient-controlled analgesia in the ESP group and control group will be compared with 24-hour morphine consumption and NRS scores at different time points. In addition, the need for rescue analgesics and patient satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* Agreed to participate in the study

Exclusion Criteria:

* Patients with infection at the injection site
* Coagulopathy Allergy to amide-type local anesthetics
* History of peripheral neuropathy
* Hepatic and/or renal failure
* Refusing the procedure
* Patients with heart disease
* Patients who have previously undergone surgery from the same area

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
opioid consumption | up to 24 hour
  The amount of morphine consumed in milligrams in the first 24 hours was determined with a patient-controlled analgesia pump.

CONTACTS AND LOCATIONS:
Overall Officials: Gökce Gişi, Principal Investigator — Kahramanmaras Sutcu Imam Universty; Gözen Öksüz, Study Director — Kahramanmaras Sutcu Imam Universty
Locations (1):
- Kahramanmaras Sutcu Imam University Hospital, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No